CLINICAL TRIAL: NCT01034644
Title: A Multinational, Multicenter, Single Visit, Exploratory Pharmacogenetic Trial and Long-term Follow-up of the PRISMS (Prevention of Relapses and Disability by Interferon Beta-1a Subcutaneously in Multiple Sclerosis) Trial
Brief Title: Pharmacogenetic Trial and Long-term Follow-up of the PRISMS Trial (PRISMS-15)
Acronym: PRISMS-15
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200136_022
Record Dates: First submitted 2009-12-09; First posted 2009-12-17 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Sclerosis
Keywords: Biomarkers; Genetic markers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood sampling for:
  Genetic markers BAbs/NAbs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PRISMS patients: This single group includes all the patients from the PRISMS study

SUMMARY:
This study, PRISMS-15 is a single visit, exploratory pharmacogenetic trial and long-term follow-up of the PRISMS (Prevention of Relapses and Disability by Interferon beta-1a Subcutaneously in Multiple Sclerosis) trial.

The aim of this trial is to provide additional data on the driving factors of IFN beta response and the long-term outcomes of Rebif® treatment.

This is a Phase IV trial involving subjects who previously participated in the PRISMS trial. To address the trial objectives, a single visit will be performed, at least 3 months after the onset of the last relapse.

ELIGIBILITY:
Inclusion Criteria:

* Was randomized in the PRISMS study
* Is willing and able to comply with the protocol
* Written informed consent given before any trial-related activities are carried out

Exclusion Criteria:

* Is unwilling or unable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group of patients coming from the PRISMS 6789 study
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The proportion of responders by group as defined by SNP (Single Nucleotide Polymorphism) markers | 1 day

SECONDARY OUTCOMES:
Current course of MS: RRMS or SPMS | 1 day
Current EDSS score | 1 day
Change in EDSS since randomization | 1 day
Immunogenicity assessment | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Verdun di Cantogno, MD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- Please call/email Central Contact for Recruiting Information in, Geneva, Switzerland

REFERENCES:
- [Derived] Sormani MP, Freedman MS, Aldridge J, Marhardt K, Kappos L, De Stefano N. MAGNIMS score predicts long-term clinical disease activity-free status and confirmed disability progression in patients treated with subcutaneous interferon beta-1a. Mult Scler Relat Disord. 2021 Apr;49:102790. doi: 10.1016/j.msard.2021.102790. Epub 2021 Jan 22. PMID 33571946